CLINICAL TRIAL: NCT00555958
Title: VBLOC™ Clinical Trial: Vagal Block for Obesity Control
Brief Title: Vagal Blocking for Obesity Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: ReShape Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBLOC; D00292-000
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Obesity
Keywords: Obesity; Bariatric surgery; Excess weight loss; Vagus nerve; Vagal blocking; VBLOC(TM) therapy
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): All study subjects will be implanted with the Maestro System, and all will receive VBLOC therapy.
  Interventions: Device: Active, implantable, intra-abdominal vagal blocking medical device

INTERVENTIONS:
Device: Active, implantable, intra-abdominal vagal blocking medical device — Intermittent, programmable, intra-abdominal vagal blocking

SUMMARY:
To determine the safety, efficacy and treatment algorithm(s) of the Maestro System in causing weight loss in obese subjects - This study will provide feasibility data regarding the potential of intra-abdominal vagus nerve down-regulation/block in the treatment of obesity.

DETAILED DESCRIPTION:
The development of innovative, safe and effective therapeutic options for the treatment of obese patients is both desirable and necessary. Gastric bypass operations are usually effective both short- and long-term but are also not available to or desired by many obese people for a variety of reasons. Gastric banding procedures are also available but have been reported to be less effective than gastric bypass operations. Diets, exercise programs and pharmaceutical agents offer short-term effectiveness for some obese patients but are all too often ineffective in the long term. The ever increasing impact of obesity on morbidity, mortality and accelerating healthcare resource utilization in most developed countries is well documented.

Activation and up-regulation of the efferent and afferent fibers of the intra-abdominal vagal nerve trunks is a pivotal physiological mechanism for food ingestion, mechanical processing, enzymatic digestion and calorie absorption. EnteroMedics' Maestro™ System is designed to take therapeutic benefit from these physiological principles by reversibly and controllably down-regulating/blocking both the anterior and posterior intra-abdominal vagal trunks in order to: (1) reduce food intake by reducing gastric volume; (2) initiate early and prolonged satiation by delaying gastric emptying; and, (3) decrease calorie absorption by down-regulating pancreatic exocrine secretion and digestion. This multi-modal mechanism is implemented in order achieve predictable and controllable loss of body weight.

This is a prospective, open-label, multi-center, clinical trial with the subjects' baseline parameters as the control. Subjects implanted laparoscopically with the Maestro System were followed from 6-months to two years.

* Implantable components: two flexible leads (including one electrode each for the anterior and posterior intra-abdominal vagal nerve trunks) that are connected to an implantable neuroregulator placed subcutaneously on the abdominal wall below the costal margin (a minimum of two or three finger widths below), or a location determined by the surgeon and consistent with device operation.
* External components:

  * For the Maestro System using a neuroregulator with an internal rechargeable battery: one mobile charger for the implanted neuroregulator, which is connected via a small, flexible cable to a cutaneous transmit coil that is positioned over the implanted neuroregulator when charging the device or determining the status of the device; a software program on a laptop computer that transmits information to the neuroregulator and uploads data from the neuroregulator, which is available to the clinician, allowing both change in treatment regimens and assessment of treatment compliance.
  * For the Maestro System using a neuroregulator with no battery: one programmable, battery-powered ambulatory controller connected via a small, flexible cable to a cutaneous transmit coil that is positioned over the implanted neuroregulator to provide power for the device; a software program on a laptop computer that transmits information to and uploads data from the controller which is available to the clinician, allowing both change in treatment regimens and assessment of treatment compliance.

The objectives of this trial are as follows:

* Determination of efficacy by quantification of excess body weight loss (EWL) at 4 and 12 weeks, and 6, 12, 24, 36, 48 and 60 months.
* Evaluation of safety through 4 and 12 weeks, and 6, 12, 24, 36, 48 and 60 months.
* Selection of effective daily treatment regimen(s).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 35-50 +/- 10% inclusive
* Failure to respond to diet/exercise program

Exclusion Criteria:

* History of gastric resection or major upper-abdominal surgery (e.g. cholycystectomy, hysterectomy acceptable)
* Current type 1 diabetes mellitus (DM) or poorly controlled type 2 DM
* Reductions of more than 10% of body weight in the previous 12 months
* Current medical condition that would make subject unfit for surgery under general anesthesia or that would be exacerbated by intentional weight loss

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2005-11; Primary Completion 2011-09 (Actual); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Excess weight loss (EWL) | 4 and 12 weeks, and 6, 12, 24, 36, 48 and 60 months
Serious Adverse Events (SAE) and Unanticipated Adverse Device Effects (UADE) | 4 and 12 weeks, and 6, 12, 24, 36, 48 and 60 months

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (2):
  - Flinders Medical Centre, Bedford Park, South Australia
  - Institute of Weight Control, Sydney
- Instituto Nacional de la Nutrición Salvador Zubiran (INNSZ), Mexico City, Mexico
- National Center for Advanced Laparoscopic Surgery, St. Olavs University Hospital, Trondheim, Norway
- University Hospital Basel, Department of Internal Medicine, Basel, Switzerland

REFERENCES:
- [Derived] Shikora S, Toouli J, Herrera MF, Kulseng B, Zulewski H, Brancatisano R, Kow L, Pantoja JP, Johnsen G, Brancatisano A, Tweden KS, Knudson MB, Billington CJ. Vagal blocking improves glycemic control and elevated blood pressure in obese subjects with type 2 diabetes mellitus. J Obes. 2013;2013:245683. doi: 10.1155/2013/245683. Epub 2013 Jul 30. PMID 23984050